CLINICAL TRIAL: NCT00120406
Title: Evaluation of the Zilver PTX Drug-Eluting Stent in the Above-the-Knee Femoropopliteal Artery
Acronym: Zilver PTX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Group Incorporated (Industry)
Collaborators: William Cook Europe (Industry); MED Institute, Incorporated (Industry); Cook Japan Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-026; PS2
Record Dates: First submitted 2005-07-11; First posted 2005-07-18 (Estimated); Results first posted 2014-08-11 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-07

CONDITIONS: Peripheral Vascular Diseases
Keywords: Peripheral Arterial Disease (PAD); Peripheral Vascular Disease; Drug-Eluting Stent; Drug-Coated Stent
MeSH Terms: conditions — Peripheral Vascular Diseases; Peripheral Arterial Disease | interventions — Angioplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Zilver® PTX™ Drug Eluting Vascular Stent
  Interventions: Device: Zilver® PTX™ Drug Eluting Vascular Stent
- 2 (Active Comparator): Angioplasty
  Interventions: Procedure: Angioplasty

INTERVENTIONS:
Device: Zilver® PTX™ Drug Eluting Vascular Stent — Stenting of the Superfemoropopliteal Artery
  Arms: 1
Procedure: Angioplasty — Angioplasty of the Superfemoropopliteal Artery
  Other Names: Balloon; PTA
  Arms: 2

SUMMARY:
The Zilver® PTX™ Drug Eluting Vascular Stent is indicated for the treatment of symptomatic vascular disease of the above-the-knee femoropopliteal artery (ranging from 4 mm to 9 mm in reference vessel diameter) for lesions up to 7 cm long. The clinical trial is stratified by lesion length. The trial will be conducted in 2 phases, with Phase 1 enrolling patients with lesions less than 7 cm long. Phase 2 of the trial will include longer lesions (up to 14 cm long) and will be initiated upon approval by the Food and Drug Administration (FDA).

DETAILED DESCRIPTION:
The Zilver® PTX™ Drug Eluting Vascular Stent is indicated for the treatment of symptomatic vascular disease of the above-the-knee femoropopliteal artery (ranging from 4 mm to 9 mm in reference vessel diameter) for lesions up to 7 cm long. The above-the-knee femoropopliteal artery is defined as the superficial femoral artery (SFA) and the region of the popliteal artery above the plane of the femoral epicondyles. The clinical trial is stratified by lesion length. The trial will be conducted in 2 phases, with Phase 1 enrolling patients with lesions less than 7 cm long. Phase 2 of the trial will include longer lesions (up to 14 cm long) and will be initiated upon approval by the FDA.

This study will include 480 patients who will receive the Zilver PTX stent or Percutaneous transluminal angioplasty (PTA) at up to 100 investigational sites. Clinical data will be captured on paper and electronic case report forms. Analyses will include evaluation of the composite event-free survival rate and the patency rate at 6- and 12-month follow-up. Event-free survival is defined as freedom from the major adverse events of death, target lesion revascularization, target limb ischemia requiring surgical intervention (bypass or amputation of toe, foot or leg), surgical repair of the target vessel (e.g., dissection requiring surgery), and from worsening of the Rutherford classification by 2 classes or to class 5 or 6. Patency will be assessed by duplex ultrasound in all patients. Patients may be randomized to one or more of the following sub-studies: IVUS and angiography at 6 months (stent patients only), angiography at 12 months, pharmacokinetic substudy (Zilver PTX patients only), or ultrasound (PTA patients only). The trial also includes provisions for patients experiencing PTA failure. These patients may be randomized to receive a Zilver PTX stent or a bare Zilver stent.

ELIGIBILITY:
Inclusion Criteria:

* Patient has signed and dated the informed consent.
* Patient has up to 2 documented stenotic or occluded atherosclerotic lesions (up ro 14 cm long) of the above-the-knee femoropopliteal artery, up to one in each limb, that meet all of the inclusion criteria and none of the exclusion criteria.
* Patient has a de novo or restenotic lesion(s) with >50% stenosis documented angiographically and no prior stent in the target lesion.
* Patient has symptoms of peripheral arterial disease classified as Rutherford Category 2 or greater.
* Patient has a resting Ankle Brachial Index (ABI) <0.9 or an abnormal exercise ABI if resting ABI is normal. Patient with incompressible arteries (ABI >1.2) must have a Toe Brachial Index (TBI) <0.8.
* Patient agrees to return for a clinical status assessment and duplex ultrasound at 6 months, 12 months, and at 2, 3, 4, and 5 years.
* Patient agrees to return for x-rays at 6 and 12 months.
* Patient agrees to return for angiography at 12 months.
* Patient agrees to be contacted by telephone at 1, 3, 9, and 18 months to assess clinical status.

Exclusion Criteria:

* Patient is pregnant or breast-feeding.
* Patient is simultaneously participating in another investigational drug or device study.
* Patient has significant stenosis or occlusion of inflow tract not successfully treated before this procedure.
* Patient has any planned surgical or interventional procedure within 30 days after the study procedure.
* Patient has had previous stenting of target vessel.
* Patient in whom antiplatelet and/or anticoagulant therapy is contraindicated.
* Patient has known hypersensitivity or contraindication to aspirin, antiplatelet medication, contrast dye, paclitaxel or nitinol and, in the opinion of the investigator, cannot be adequately premedicated.
* Patient lacks at least one patent vessel of runoff with <50% stenosis throughout its course.
* Patient has untreated angiographically-evident thrombus in the target lesion.

[Additional criteria may apply.]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 474 (Actual)
Dates: Start 2005-03; Primary Completion 2009-10 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dake, M.D., Principal Investigator — Stanford University
Locations (52):
- United States (44):
  - El Camino Hospital, Mountain View, California
  - Tri-City Medical Center, Oceanside, California
  - Stanford University Hospital and Clinics, Stanford, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - JFK Memorial Center, Atlantis, Florida
  - University of Florida, Gainesville, Florida
  - Memorial -- Jacksonville, Jacksonville, Florida
  - Baptist Cardiac & Vascular Institute, Miami, Florida
  - Orlando Regional Medical Center, Orlando, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Prairie Heart, Springfield, Illinois
  - St. Vincent Hospital, Indianapolis, Indiana
  - The Care Group, Indianapolis, Indiana
  - Christus St. Patrick Hospital, Lake Charles, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Bayview Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Michigan Vascular Research Center, Flint, Michigan
  - William Beaumont, Royal Oak, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - St. Luke's Hospital Kansas, Kansas City, Missouri
  - NYU Medical Center, New York, New York
  - St. Luke's Roosevelt Hospital Center, New York, New York
  - New York Presbyterian Hospital, New York, New York
  - Lenox Hill, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Good Samaritan Hospital, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - MidWest Cardiology Research Foundation, Columbus, Ohio
  - EMH Regional Medical Center, Elyria, Ohio
  - University of Toledo University Medical Center, Toledo, Ohio
  - Pinnacle Health Harrisburg, Harrisburg, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - South Carolina Heart Center, Columbia, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Methodist Hospital, Houston, Texas
  - Peripheral Vascular Associates (PVA), San Antonio, Texas
  - LDS, Murray, Utah
  - University of Virginia Medical Center, Charlottesville, Virginia
  - St. Luke's Hospital, Milwaukee, Wisconsin
- Germany (4):
  - Herz-Zentrum, Bad Krozingen
  - Gemeinschaftspraxis, Leipzig
  - Heart Center Leipzig, Angiology, Leipzig
  - Universitatsklinikum Magdeburg, Magdeburg
- Japan (4):
  - Kokura Memorial Hospital, Kitakyushu, Fukuoka
  - The Jikei University Hospital, Nishi-Shinbashi, Minato-ku
  - Kyoto University Hospital, Kyoto
  - Nara Medical University, Nara

REFERENCES:
- [Derived] Dake MD, Fanelli F, Lottes AE, O'Leary EE, Reichert H, Jiang X, Fu W, Iida O, Zen K, Schermerhorn M, Zeller T, Ansel GM. Prediction Model for Freedom from TLR from a Multi-study Analysis of Long-Term Results with the Zilver PTX Drug-Eluting Peripheral Stent. Cardiovasc Intervent Radiol. 2021 Feb;44(2):196-206. doi: 10.1007/s00270-020-02648-6. Epub 2020 Oct 6. PMID 33025243
- [Derived] Dake MD, Ansel GM, Jaff MR, Ohki T, Saxon RR, Smouse HB, Machan LS, Snyder SA, O'Leary EE, Ragheb AO, Zeller T; Zilver PTX Investigators. Durable Clinical Effectiveness With Paclitaxel-Eluting Stents in the Femoropopliteal Artery: 5-Year Results of the Zilver PTX Randomized Trial. Circulation. 2016 Apr 12;133(15):1472-83; discussion 1483. doi: 10.1161/CIRCULATIONAHA.115.016900. Epub 2016 Mar 11. PMID 26969758
- [Derived] Ohki T, Yokoi H, Kichikawa K, Kimura T, Snyder SA, Ragheb AO, O'Leary EE, Jaff MR, Ansel GM, Dake MD. Two-year analysis of the Japanese cohort from the Zilver PTX randomized controlled trial supports the validity of multinational clinical trials. J Endovasc Ther. 2014 Oct;21(5):644-53. doi: 10.1583/14-4753.1. PMID 25290792
- [Derived] Dake MD, Ansel GM, Jaff MR, Ohki T, Saxon RR, Smouse HB, Snyder SA, O'Leary EE, Tepe G, Scheinert D, Zeller T; Zilver PTX Investigators. Sustained safety and effectiveness of paclitaxel-eluting stents for femoropopliteal lesions: 2-year follow-up from the Zilver PTX randomized and single-arm clinical studies. J Am Coll Cardiol. 2013 Jun 18;61(24):2417-2427. doi: 10.1016/j.jacc.2013.03.034. Epub 2013 Apr 10. PMID 23583245
- [Derived] Dake MD, Ansel GM, Jaff MR, Ohki T, Saxon RR, Smouse HB, Zeller T, Roubin GS, Burket MW, Khatib Y, Snyder SA, Ragheb AO, White JK, Machan LS; Zilver PTX Investigators. Paclitaxel-eluting stents show superiority to balloon angioplasty and bare metal stents in femoropopliteal disease: twelve-month Zilver PTX randomized study results. Circ Cardiovasc Interv. 2011 Oct 1;4(5):495-504. doi: 10.1161/CIRCINTERVENTIONS.111.962324. Epub 2011 Sep 27. PMID 21953370

RESULTS

PARTICIPANT FLOW:
Groups:
- Zilver PTX: Zilver® PTX™ Drug Eluting Vascular Stent
- PTA (Control): Percutaneous balloon angioplasty
Period: Overall Study
Arm/Group | Zilver PTX | PTA (Control)
Started | 236 | 238
Completed | 217 | 222
Not Completed | 19 | 16
Not completed — Death | 9 | 4
Not completed — Withdrawal by Subject | 5 | 7
Not completed — Lost to Follow-up | 5 | 2
Not completed — received non-study stent | 0 | 2
Not completed — patient moved but has not withdrawn | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zilver PTX | PTA (Control) | Total
Number analyzed (Participants) | 236 | 238 | 474
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.9 (9.6) | 67.7 (10.6) | 67.8 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 86 | 167
  Male | 155 | 152 | 307
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body mass index
  kg/m^2 | 28.4 (5.3) | 28.2 (5.6) | 28.3 (5.4)
Diabetes [Number; unit: participants]
  Patients with diabetes | 117 | 100 | 217
  Patients without diabetes | 119 | 138 | 257
Hypercholesterolemia [Number; unit: participants]
  Patients with hypercholesterolemia | 180 | 166 | 346
  Patients without hypercholesterolemia | 56 | 72 | 128
Hypertension [Number; unit: participants]
  Patients with hypertension | 210 | 194 | 404
  Patients without hypertension | 26 | 44 | 70
Smoking status [Number; unit: participants]
  Never smoked | 32 | 37 | 69
  Quit | 131 | 123 | 254
  Still smokes | 73 | 77 | 150
  Unknown | 0 | 1 | 1
Stenosed lesion length [Mean (Standard Deviation); unit: mm] — Region with > 20% diameter stenosis (242 lesions in the PTX group and 248 lesions in the PTA group)
  mm | 54.6 (40.7) | 53.2 (40.3) | 53.9 (40.5)
Normal-to-normal Lesion length [Mean (Standard Deviation); unit: mm] — Site reported diseased lesion length (246 lesions in the PTX group and 251 lesions in the PTA group)
  mm | 66.4 (38.9) | 63.2 (40.5) | 64.8 (39.7)
Percent diameter stenosis [Mean (Standard Deviation); unit: percent of proximal ref. vessel diameter] — 242 lesions in the PTX group and 249 lesions in the PTA group
  percent of proximal ref. vessel diameter | 79.8 (17) | 78.4 (17.1) | 79.1 (17)
Total Occlusion [Number; unit: lesions]
  Lesions with total occlusion | 79 | 68 | 147
  Lesions without total occlusion | 162 | 180 | 342
Calcification [Number; unit: lesions]
  None | 4 | 12 | 16
  Little | 62 | 95 | 157
  Moderate | 85 | 55 | 140
  Severe | 90 | 87 | 177

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival Rate
Description: Event-free survival is defined as freedom from the major adverse events of death, target lesion revascularization, target limb ischemia requiring surgical intervention (bypass or amputation of toe, foot or leg), surgical repair of the target vessel (e.g., dissection requiring surgery), and from worsening of the Rutherford classification by 2 classes or to class 5 or 6.
  Participant flow is based on initial randomization of Zilver PTX or PTA (Percutaneous balloon angioplasty), and Event-free survival is based on Per-Protocol analysis where only patients who were treated according to their initial randomization are counted.
Time Frame: 12 months
Measure: Number; unit: Percentage of participants
Arm/Group | Zilver PTX | PTA (Control)
Number analyzed (Participants) | 235 | 236
Percentage of participants | 90.4 | 83.9
Statistical Analysis 1: Comparison: Zilver PTX vs PTA (Control); Test type: Non-Inferiority or Equivalence — Non-inferiority margin is 10%; p < 0.01, z-test, one-sided — P-value has been adjusted for multiplicity

2. Primary Outcome: Primary Patency
Description: Primary patency is defined as a Peak systolic velocity (PSV) ratio < 2.0 or angiographic percent diameter stenosis < 50%.
Time Frame: 12 months
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Lesions
Arm/Group | Zilver PTX | PTA (Control)
Number analyzed (Participants) | 236 | 238
Number analyzed (Lesions) | 246 | 251
Percentage of participants | 82.7 | 32.7
Statistical Analysis 1: Comparison: Zilver PTX vs PTA (Control); Test type: Superiority or Other; p < 0.01, Generalized estimating equation (GEE) — P-value has been adjusted for multiplicity

ADVERSE EVENTS:
Time Frame: 12 months
Description: Participant flow is based on initial randomization of Zilver PTX or PTA (Percutaneous balloon angioplasty), and adverse events are based on Per-Protocol analysis where only patients who were treated according to their initial randomization are counted.
Arm/Group | Zilver PTX | PTA (Control)
Serious Adverse Events (participants affected / at risk) | 21/235 | 37/236
Other Adverse Events (participants affected / at risk) | 81/235 | 72/236
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zilver PTX (N=235) | PTA (Control) (N=236)
Clinically-driven TLR (Target Lesion Revascularization) (Vascular disorders) | 21 (21) | 36 (36)
Worsening of Rutherford classification by 2 classes or to a class 5 or 6 (Vascular disorders) | 0 (0) | 2 (2)
Amputation (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zilver PTX (N=235) | PTA (Control) (N=236)
Pneumonia requiring antibiotics (Respiratory, thoracic and mediastinal disorders) | 12 (14) | 5 (6)
Post-procedure percutaneous intervention (e.g., PTA and/or stent) to the study vessel (Vascular disorders) | 13 (14) | 19 (22)
Post-procedure percutaneous intervention (e.g., PTA and/or stent) to another vessel (Vascular disorders) | 50 (62) | 40 (52)
Worsened claudication/rest pain (Vascular disorders) | 10 (12) | 16 (21)
Post-procedure transfusion (Vascular disorders) | 13 (13) | 10 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days